CLINICAL TRIAL: NCT07355569
Title: Sending SMS Notification Prior to a Scheduled Screening Appointment in BreastScreen Norway - the Effect on Attendance
Brief Title: The Effect on Attendance of an SMS Notification Prior to a Scheduled Screening Appointment in BreastScreen Norway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 5158-5158
Record Dates: First submitted 2026-01-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Attendance; Breast Cancer Screening
Keywords: breast cancer screening; SMS notification; attendance

STUDY DESIGN:
Intervention Model Description: Simple 1:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The intervention was an SMS notification sent before the scheduled appointment for mammographic screening. Women in the study group was linked to the Common Contact Register in Norway (CCRN) to obtain phone numbers for sending SMS notification prior to the scheduled appointment. Phone numbers are registered in CCRN when users log into public online services through an electronic ID. Inclusion in this registry is voluntary. The personal identification number of the women in the study group was used to obtain their phone number.
  In study group 1 women were linked to the CCRN and those registered were sent an SMS notification three days prior to the scheduled routine screening appointment during January-March 2025. Women in study group 2 were sent an SMS notification two days prior to the scheduled routine screening appointment during April-June 2025.
  Interventions: Other: SMS notification
- Control group (No Intervention): Women in the control group did not receive any SMS notification before the scheduled appointment to mammographic screening. The women in the control group were not linked to the NCCR and were not available or sent an SMS notification during the study periods, January-March 2025 (control group 1) and women who were not sent an SMS notification during April-June 2025 (control group 2).

INTERVENTIONS:
Other: SMS notification — Available in the NCCR and sent an SMS notification three or two days prior to a scheduled screening appointment
  Arms: Study group

SUMMARY:
This study has been designed as a randomized controlled trial including women invited to a national screening program for breast cancer in Norway, BreastScreen Norway in 2025. The program invites women aged 50-69 to biennial screening mammography. The study includes two substudies with the intervention of sending an SMS notification three days prior to the screening appointment in the first substudy and two days prior to the screening appointment in second study. The comparison is made between the study groups, where women are sent an SMS notification two or three days prior to their scheduled screening appointment and the control groups where women will not be sent an SMS notification about a scheduled screening appointment.

ELIGIBILITY:
Inclusion Criteria:

* women invited to BreastScreen Norway residing in the South-Eastern, Central, and Northern Norway Regional Health Authorities

Exclusion Criteria:

* no

Ages: 50 Years to 71 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133770 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Screening attendance | Three months (180 days) after scheduled date for a screening examination following a routine invitation or three months (180 days) after a reminder was posted.
  Attendance after a routine or reminder invitation, with and without an SMS notification

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian Institute of Public Health, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No
Research data, including participant data used can only be requested from https://helsedata.no/, given the legal basis in Articles 6 and 9 of the GDPR and that the processing is in accordance with Article 5 of the GDPR, as well as Norwegian legislation.